CLINICAL TRIAL: NCT00702325
Title: A 12-wk, Rand., Double-blind, Double Dummy, Multi-ctr., Phase IV Study Comparing Efficacy and Safety of SYMBICORT® pMDI 160/4.5 ug x 2 Actuations Twice Daily Versus Pulmicort® (Budesonide Inhalation Powder DPI) 180 ug x 2 Inhalations Twice Daily, in Adult and Adolescent African American Subjects With Asthma
Brief Title: Phase4/Symbicort® Versus Pulmicort Flexhaler® in African Americans
Acronym: Titan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D589BL00003
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Results first posted 2012-11-09 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-10

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; Formoterol Fumarate; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Budesonide / formoterol fumarate (SYMBICORT)
- 2 (Active Comparator)
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Budesonide / formoterol fumarate (SYMBICORT) — 160/4.5 μg x 2 actuations twice daily (bid)
  Other Names: SYMBICORT
  Arms: 1
Drug: Budesonide — inhalation powder 180 μg x 2 inhalations bid (PULMICORT)
  Other Names: PULMICORT
  Arms: 2

SUMMARY:
To compare the efficacy of SYMBICORT® pMDI 160/4.5 μg x 2 actuations twice daily (bid) to that of budesonide inhalation powder DPI 180 μg x 2 inhalations bid, in African American(self-reported) subjects with inhaled corticosteroid (ICS) dependent asthma.

ELIGIBILITY:
Inclusion Criteria:

* African American (self-reported)
* Documented clinical diagnosis of asthma as defined by the American Thoracic Society (ATS) for at least 6 months prior to Visit 2 and be in stable condition.
* FEV1, measured ≥6 hours after the last dose of short-acting β2-agonist and at least 48 hours after LABA, of 45%-85%, inclusive, of predicted normal.

Exclusion Criteria:

* Has been hospitalized at least once for an asthma related condition during the 6 months prior to Visit 2, or has required emergency treatment due to an asthma related condition more than once in the 3 months prior to Visit 2.
* Has required treatment with systemic corticosteroids (eg, oral, parenteral, ocular, or rectal) for any reason within the 30 days prior to Visit 2.
* Has a respiratory infection or other viral/bacterial illness, or is recovering from such an illness at the time of Visit 3 that, in the Investigator's opinion, will interfere with the subject's lung function and/or ability to perform spirometry

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ubaldo Martin, MD, Study Director — AstraZeneca; Tomas LG Andersson, Study Director — AstraZeneca
Locations (57):
- United States (57):
  - Research Site, Pell City, Alabama
  - Research Site, Bentonville, Arkansas
  - Research Site, Hot Springs, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Malvern, Arkansas
  - Research Site, Huntington Park, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Los Angles, California
  - Research Site, Orange, California
  - Research Site, Rolling Hills Estates, California
  - Research Site, Centennial, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Waterbury, Connecticut
  - Research Site, Inverness, Florida
  - Research Site, Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, Tampa, Florida
  - Research Site, Alpharetta, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Lithia Springs, Georgia
  - Research Site, Lovejoy, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Hagerstown, Maryland
  - Research Site, Lanham, Maryland
  - Research Site, Largo, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Flint, Michigan
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Skillman, New Jersey
  - Research Site, New York, New York
  - Research Site, North Syracuse, New York
  - Research Site, Durham, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Portland, Oregon
  - Research Site, Blue Bell, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, McKinney, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Waco, Texas
  - Research Site, Emporia, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Murphy KR, Uryniak T, Martin UJ, Zangrilli J. The effect of budesonide/formoterol pressurized metered-dose inhaler on predefined criteria for worsening asthma in four different patient populations with asthma. Drugs R D. 2012 Mar 1;12(1):9-14. doi: 10.2165/11630600-000000000-00000. PMID 22329608

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrolled on 05 June 2008, last participant last visit on 10 September 2009.
Pre-assignment Details: 10 subjects were excluded from the FAS: 9 who received the incorrect study medication and 1 who was randomized to receive SYMBICORT pMDI, but never received study medication.
  Therefore, 153 subjects (from 156 randomized to Symbicort) and 148 (from 155 randomized to Budesonide) were included in the FAS used to present baseline characteristics.
Groups:
- Symbicort: Symbicort pressurized metered dose inhaler (pMDI) 160/4.5 mcg x 2 actuations, twice daily.
- Budesonide: Budesonide inhalation dry powder inhaler (DPI) 180 mcg x 2 inhalations, twice daily.
Period: Overall Study
Arm/Group | Symbicort | Budesonide
Started | 156 (Randomized) | 155 (Randomized)
Completed | 118 (Completed participants based on randomized population (156) minus discontinued participants (38).) | 102 (Completed participants based on randomized population (155) minus discontinued participants (53).)
Not Completed | 38 | 53
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 7 | 7
Not completed — Lost to Follow-up | 3 | 4
Not completed — Incorrect enrollment | 5 | 7
Not completed — Developed study discontinuation criteria | 18 | 28
Not completed — Severe noncompliance to protocol | 3 | 3
Not completed — Termination due to lab results | 1 | 0
Not completed — Didn't follow study medication dosage | 0 | 2
Not completed — Withdrew consent | 0 | 1
Not completed — Incorrectly Discontinued | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Symbicort | Budesonide | Total
Number analyzed (Participants) | 153 | 148 | 301
Age Continuous [Mean (Standard Deviation); unit: Years] | 38.6 (13.8) | 39.8 (15.4) | 39.2 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 87 | 196
  Male | 44 | 61 | 105

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pre-dose Forced Expiratory Volume in 1 Second (FEV1) Averaged Over Treatment Period
Description: Mean change from baseline (Visit 3) value to average value recorded at visits during treatment period
Time Frame: Baseline to 12 weeks
Population: Full analysis set (FAS) was performed and was based on data from all subjects who were randomized, took at least 1 dose of study medication, and contributed sufficient data for calculation of this outcome Measure.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 150 | 143
Liters | 0.16 (0.31) | 0.07 (0.26)

2. Secondary Outcome: Change From Baseline in Morning Peak Expiratory Flow (AM PEF) Averaged Over the Treatment Period
Description: Mean change from baseline (Visit 3) value to average value recorded at visits during treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 149 | 139
Liters/minute | 25.34 (43.70) | 7.53 (32.41)

3. Secondary Outcome: Change From Baseline in Evening Peak Expiratory Flow (PM PEF) Averaged Over the Treatment Period
Description: Mean change from baseline (Visit 3) value to average value recorded at visits during treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 149 | 141
Liters/minute | 21.61 (40.75) | 7.67 (48.97)

4. Secondary Outcome: Change From Baseline in Pre-dose Forced Vital Capacity (FVC) Averaged Over the Treatment Period
Description: Mean change from baseline (Visit 3) value to average value recorded at visits during treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 150 | 143
Liters | 0.14 (0.32) | 0.07 (0.27)

5. Secondary Outcome: Change From Baseline in Pre-dose Forced Expiratory Flow (FEF 25-75%) Averaged Over the Treatment Period
Description: Mean change of the FEF (25-75%) value at the baseline (Visit 3) compared to average value of the FEF (25-75%) recorded at visits during treatment period (to week 12). The mean change was calculated.
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters/second
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 150 | 143
Liters/second | 0.21 (0.47) | 0.12 (0.47)

6. Secondary Outcome: Number of First Predefined Asthma Events by Inhaled Corticosteroid (ICS) Dose at Entry
Description: Total number of participants with any first predefined asthma event (decrease in FEV1 ≥ 20%,or to <40% of predicted normal value,12 puffs of albuterol pMDI per day on 3 or more days, decrease in morning PEF ≥ 20% on 3 or more days, use of rescue medication for 2 or more nights, emergency treatment, hospitalization, use of other asthma medication)
Time Frame: 12 weeks
Measure: Number; unit: Participants
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 153 | 148
Participants | 57 | 67

7. Secondary Outcome: Number of Withdrawals Due to a Predefined Asthma Event
Description: Total number of participants who withdrew due to a predefined asthma event (decrease in FEV1 ≥ 20%,or to <40% of predicted normal value,12 puffs of albuterol pMDI per day on 3 or more days, decrease in morning PEF ≥ 20% on 3 or more days, use of rescue medication for 2 or more nights, emergency treatment, hospitalization, use of other asthma meds)
Time Frame: 12 weeks
Measure: Number; unit: Participants
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 153 | 148
Participants | 18 | 28

8. Secondary Outcome: Change From Baseline in Total Average Daily Asthma Symptom Score Averaged Over the Treatment Period
Description: Diary assessment of total asthma symptoms score (treatment average) by Inhaled Corticosteroid (ICS) dose at entry. Asthma symptoms are cough, wheeze and shortness of breath. Each symptom is usually rated from 0-3: 0-no symptoms, 1-mild, 2-moderate and 3-severe. Change from baseline (Visit 3) mean value to average value recorded at visits during treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 149 | 142
Scores on a scale | -0.35 (0.42) | -0.23 (0.40)

9. Secondary Outcome: Change From Baseline in Nighttime Asthma Symptom Score Averaged Over the Treatment Period
Description: Diary assessment of nighttime asthma symptoms score (treatment average) by ICS dose at entry. Asthma symptoms are cough, wheeze and shortness of breath. Each symptom is usually rated from 0-3: 0-no symptoms, 1-mild, 2-moderate and 3-severe. Change from baseline (Visit 3) mean value to average value recorded at visits during treatment period; full analysis set (FAS)
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 151 | 146
Scores on a scale | -0.38 (0.47) | -0.26 (0.42)

10. Secondary Outcome: Change From Baseline in Daytime Asthma Symptom Score Averaged Over the Treatment Period
Description: Diary assessment of daytime asthma symptoms score (treatment average) by ICS dose at entry. Asthma symptoms are cough, wheeze and shortness of breath. Each symptom is usually rated from 0-3: 0-no symptoms, 1-mild, 2-moderate and 3-severe. Change from baseline (Visit 3) mean value to average value recorded at visits during treatment period; full analysis set (FAS)
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 150 | 143
Scores on a scale | -0.33 (0.45) | -0.24 (0.45)

11. Secondary Outcome: Change From Baseline in Awakening-free Nights Averaged Over the Treatment Period
Description: Diary assessment of number of nights free from awakenings due to asthma; mean change from baseline (Visit 3) value to average value recorded at visits during treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of nights
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 150 | 143
Number of nights | 17.51 (26.51) | 11.85 (25.92)

12. Secondary Outcome: Change From Baseline to the Average in Total Rescue Medication Use Averaged Over the Treatment Period
Description: Diary assessment of total daily puffs of rescue medication used for asthma symptoms relief; mean change from baseline (Visit 3) value to average value recorded at visits during treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Puffs/day
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 150 | 144
Puffs/day | -1.27 (1.81) | -0.62 (1.68)

13. Secondary Outcome: Change From Baseline to the Average in Nighttime Rescue Medication Use Averaged Over the Treatment Period
Description: Diary assessment of total nighttime puffs of rescue medication used for asthma symptoms relief; mean change from baseline (Visit 3) value to average value recorded at visits during treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Puffs/day
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 150 | 144
Puffs/day | -0.79 (1.07) | -0.35 (0.93)

14. Secondary Outcome: Change From Baseline to the Average in Daytime Medication Use Averaged Over the Treatment Period
Description: Diary assessment of total daytime puffs of rescue medication used for asthma symptoms relief; mean change from baseline (Visit 3) value to average value recorded at visits during treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Puffs/day
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 150 | 144
Puffs/day | -0.48 (0.93) | -0.27 (0.92)

15. Secondary Outcome: Change From Baseline to the Average in Rescue Medication-free Days Averaged Over the Treatment Period
Description: Diary assessment of total (percent) days free from rescue medication use for asthma symptoms relief; mean change from baseline (Visit 3) value to average value recorded at visits during treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 150 | 144
percentage of days | 29.31 (34.13) | 17.70 (35.39)

16. Secondary Outcome: Change From Baseline in Asthma Symptom-free Days Averaged Over the Treatment Period
Description: Diary assessment of number (percent) of days free from asthma symptoms by ICS dose at entry; mean change from baseline (Visit 3) value to average value recorded at visits during treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 151 | 146
percentage of days | 23.99 (29.82) | 17.55 (28.58)

17. Secondary Outcome: Change From Baseline to the Average for Asthma-control Days Averaged Over the Treatment Period
Description: Diary assessment of number (percent) of asthma-control days (defined as days that were free of symptoms and nighttime and daytime rescue medication use); mean change from baseline (Visit 3) value to average value recorded at visits during treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 151 | 147
percentage of days | 21.89 (29.48) | 15.12 (26.80)

18. Secondary Outcome: Perception of Onset of Medication Effect at Last Week of Treatment Assessed by Number of Participants Who Agreed With Item 2 on the Onset of Effect Questionnaire (OEQ)
Description: Diary assessment of participants age 12 years and older and 18 years and older who agreed with OEQ Item 2 at last week of treatment - During the past week, you could feel your medication begin to work right away
Time Frame: 12 week
Measure: Number; unit: Participants
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 144 | 136
Participants
  12 years and older | 123 | 112
  18 years and older | 109 | 95

19. Secondary Outcome: Change From Baseline to End of Treatment in Overall Score on the Asthma Quality of Life Questionnaire-Standardized (AQLQ[S])
Description: Mean change in overall score at end of treatment for participants age 17 years and older (scores ranged from 1 to 7, with higher scores indicating better quality of life); mean change from baseline (Visit 3) value to average value recorded at visits during treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 125 | 123
Scores on a scale | 0.55 (0.96) | 0.33 (1.07)

20. Secondary Outcome: Proportion of Participants Who Reported on the Asthma Control Test (ACT) That Their Asthma Was Controlled at the Last Week of Treatment
Description: There are 5 questions in the survey, and each question has 5 responses (total score for each question can range from 1 to 5). To score the survey, responses to the 5 questions are added to yield a total score that ranges from 5 (poor control of asthma control) to 25 (complete control of asthma). Score of 20 or higher was indicative of well-controlled asthma.
Time Frame: 12 weeks
Measure: Number; unit: Proportion of Participants
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 143 | 139
Proportion of Participants | 0.524 | 0.518

21. Secondary Outcome: Change From Baseline to Last Week of Treatment in Scores on the Asthma Impact Survey (AIS)
Description: There are 6 questions in the survey, and each question has 5 responses (total score for each question can range from 6 to 13). Responses to the 6 questions were added to yield a total score that ranged from 36 to 78. Scoring is based on a norm-based method. Higher AIS scores indicated more asthma impact and poorer quality of life; mean change from baseline (Visit 3) value to average value recorded at visits during treatment period.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 128 | 124
Scores on a scale | -4.05 (6.79) | -2.72 (9.75)

22. Secondary Outcome: Perception of Onset of Medication Effect at Last Week of Treatment Assessed by Number of Participants Who Agreed With Item 5 on the Onset of Effect Questionnaire (OEQ)
Description: Diary assessment of participants age 12 years and older and 18 years and older who agreed with OEQ Item 5 at last week of treatment - During the past week, you were satisfied with how quickly you felt your study medication began to work.
Time Frame: 12 week
Measure: Number; unit: Participants
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 144 | 136
Participants
  12 years and older | 112 | 99
  18 years and older | 100 | 81

23. Secondary Outcome: Perception of Onset of Medication Effect at First Week of Treatment Assessed by Number of Participants Who Agreed With Item 2 on the Onset of Effect Questionnaire (OEQ)
Description: Diary assessment of participants age 12 years and older and 18 years and older who agreed with OEQ Item 2 at first week of treatment - During the past week, you could feel your medication begin to work right away
Time Frame: 1 week
Measure: Number; unit: Participants
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 256 | 234
Participants
  12 years and older | 113 | 95
  18 years and older | 101 | 81

24. Secondary Outcome: Perception of Onset of Medication Effect at First Week of Treatment Assessed by Number of Participants Who Agreed With Item 5 on the Onset of Effect Questionnaire (OEQ)
Description: Diary assessment of participants age 12 years and older and 18 years and older who agreed with OEQ Item 5 at first week of treatment - During the past week, you were satisfied with how quickly you felt your study medication began to work.
Time Frame: 1 week
Measure: Number; unit: Participants
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 256 | 234
Participants
  12 years and older | 96 | 83
  18 years and older | 86 | 70

ADVERSE EVENTS:
Arm/Group | Symbicort | Budesonide
Serious Adverse Events (participants affected / at risk) | 1/156 | 2/155
Other Adverse Events (participants affected / at risk) | 18/156 | 12/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort (N=156) | Budesonide (N=155)
Pyrexia (General disorders) | 0 | 1
Ovarian Cyst Ruptured (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort (N=156) | Budesonide (N=155)
Nasopharyngitis (Infections and infestations) | 8 | 4
Headache (Nervous system disorders) | 10 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If Sponsor does not publish within 2 years after study completion, PI is permitted to publish, with confidential information removed from manuscript. Sponsor will have opportunity to review and approve publication at least 60 days pior to being submitted/disclosed. Sponsor can request, in writing, an additional 90 day embargo.